CLINICAL TRIAL: NCT06344364
Title: Epidemiologic Liver Outcomes Retrospective Study to Confirm The Prognostic Value of the FibroNest Digital Pathology Fibrosis Biomarker (Ph-FCS) in Patients With MASLD (DPAILO-1)
Brief Title: Digital Pathology and AI for Liver Outcomes in MASLD
Acronym: DPAILO-1
Status: Not yet recruiting | Type: Observational
Sponsor: PharmaNest, Inc (Industry)
Collaborators: Chinese University of Hong Kong (Other); University of Seville (Other); Fundacio Clinic Barcelona (Other); Sorbonne University (Other)
Responsible Party: Sponsor
Other Study IDs: PHN 1-080-23
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: NAFLD; MAFLD; digital pathology; artificial intelligence; fibrosis score; liver disease; hepatic decompensation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-Liver Related Event: Absence of any of the liver events described in the second group in the patient clinical follow-up.
  Interventions: Diagnostic Test: Digital Pathology FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS)
- Liver Related Event: Liver-related events include liver-related death, hepatic decompensation events (variceal hemorrhage, ascites, hepatic encephalopathy), and hepatocellular carcinoma.
  Interventions: Diagnostic Test: Digital Pathology FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS)

INTERVENTIONS:
Diagnostic Test: Digital Pathology FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS) — Biomarker name: FibroNest Phenotypic Fibrosis Composite Score Acronym: FibroNest Ph-FCS Type of Biomarker: Histologic based, Digital, Quantitative Image Analysis, Imaging modality Definition: A quantitative, normalized (no unit) and continuous composite score that aggregates quantitative histological features of fibrosis severity measured by high resolution quantitative image analysis.

SUMMARY:
The aim of this multi-center, retrospective epidemiologic study is to confirm the prognostic performance of the Digital Pathology (DP) FibroNest Phenotypic Fibrosis Composite Score (Ph-FCS), derived from standard digital pathology liver biopsy images, in predicting clinical hepatic decompensation events in patients with metabolic dysfunction-associated steatohepatitis (MASH).

DETAILED DESCRIPTION:
MASH, or metabolic dysfunction-associated steatohepatitis, presents histological liver changes resembling those caused by alcohol abuse, but in the absence of alcohol intake. Common among adults with conditions like obesity and type-2 diabetes, MASH, especially its severe form, is anticipated to become a leading cause of end-stage liver disease.

Currently lacking approved treatments, MASH poses a significant burden on liver health and transplantation. Diagnosis and assessment rely on subjective histological review, prone to variability and limitations in detecting subtle changes. Consequently, there's an urgent need for accurate, continuous histological biomarkers.

The FibroNest Ph-FCS offers a promising solution, utilizing high resolution digital pathology and sophisticated algorithmic methods for sensitive and reproducible fibrosis severity assessment and prediction of clinical events. In a 2003 proof of concept retrospective study on 400 patients, its prognostic performance was excellent.

In this proposed multi-center retrospective study, we aim to confirm the Ph-FCS's prognostic value on a large cohort of 1,700 MASLD patients. We will also compare the prognostic performance of the Ph-FCS with the prognostic performance of the NASH-CR Fibrosis stages, and with non-invasive biomarkers like Fib-4 and elastography/Fibroscan, also collected retrospectively from the point of initial diagnosis.

This study seeks to:

(i) Confirm Ph-FCS's prognostic utility on a large scale.

(ii) Compare biopsy-based Ph-FCS with NASH-CRN F Stages

(iii) Compare biopsy-based Ph-FCS with non-invasive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Adult pts ( >=18 years old) with MASLD defined histologically.
* Liver biopsy with fibrosis stains available for digitization or already digitized.
* Clinical follow-up >1 year available recording liver-related outcomes either through hospitalization ICD-10 codes or through clinical observation

Exclusion Criteria:

* Liver diseases other than MASLD Note: no exclusion based on bariatric surgery, significant weight loss or enrollment in NASH clinical studies, but data is collected for data analysis / competing effects (see data analysis plan)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pts ( >=18 years old) with MASLD defined histologically with >1 year of clinical follow up and available recording liver-related outcomes either through hospitalization ICD-10 codes or through clinical observation.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Performance of Hepatic Decompensation Event predictive value of the FibroNest Ph-FCS | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of the FibroNest Ph-FCS, as a prognostic/diagnostic biomarker for liver related events in patients with MASH.

SECONDARY OUTCOMES:
Performance of Hepatic Decompensation Event predictive value of the NASH-CRN Fibrosis Stage, a biopsy-based score for fibrosis severity | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of NASH-CRN F stage, as a biopsy-based prognostic/diagnostic biomarker for Hepatic Decompensation Events in patients with MASH.
Performance of Hepatic Decompensation Event predictive value of the FIB-4 biomarker, a non-invasive test | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of FIB-4, as a prognostic/diagnostic biomarker for Hepatic Decompensation Events in patients with MASH.
Performance of Hepatic Decompensation Event predictive value of the elastography (Fibroscan) biomarker, a non-invasive test | Time-to-event analysis between 2 and 10 years
  Area under Receiver Operating Characteristic Curve (AUROC) of elastography, as a prognostic/diagnostic biomarker for Hepatic Decompensation Events in patients with MASH.

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Ratziu, MD, PhD, Principal Investigator — Sorbonne University
Locations (3):
- The Chinese University of Hong Kong, Shatin, Hong Kong
- Spain (2):
  - Fundació de Recerca Clinic Barcelona, Barcelona
  - University of Seville, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanyal AJ, Van Natta ML, Clark J, Neuschwander-Tetri BA, Diehl A, Dasarathy S, Loomba R, Chalasani N, Kowdley K, Hameed B, Wilson LA, Yates KP, Belt P, Lazo M, Kleiner DE, Behling C, Tonascia J; NASH Clinical Research Network (CRN). Prospective Study of Outcomes in Adults with Nonalcoholic Fatty Liver Disease. N Engl J Med. 2021 Oct 21;385(17):1559-1569. doi: 10.1056/NEJMoa2029349. PMID 34670043
- [Background] Kendall TJ, Jimenez-Ramos M, Turner F, Ramachandran P, Minnier J, McColgan MD, Alam M, Ellis H, Dunbar DR, Kohnen G, Konanahalli P, Oien KA, Bandiera L, Menolascina F, Juncker-Jensen A, Alexander D, Mayor C, Guha IN, Fallowfield JA. An integrated gene-to-outcome multimodal database for metabolic dysfunction-associated steatotic liver disease. Nat Med. 2023 Nov;29(11):2939-2953. doi: 10.1038/s41591-023-02602-2. Epub 2023 Oct 30. PMID 37903863
- [Background] Ratziu V, Chen L, Petitjean L. et al. Novel Artificial Intelligence-Assisted Digital Pathology Quantitative Image Analysis Predicts the occurrence of Liver-related Clinical Events in the Multicentric, European, Hepatic Outcomes and Survival Fatty Liver Registry (HITSURFR) Study. Hepatology. 78(S1) S1-S2154 2084-A